CLINICAL TRIAL: NCT04264143
Title: A Phase I Study Examining the Feasibility of Intermittent Convection-Enhanced Delivery (CED) of MTX110 for the Treatment of Children With Newly Diagnosed Diffuse Midline Gliomas
Brief Title: CED of MTX110 Newly Diagnosed Diffuse Midline Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luca Szalontay (Other)
Collaborators: Midatech Pharma US Inc. (Industry)
Responsible Party: Sponsor-Investigator, Luca Szalontay, Herbert and Florence Irving Associate Professor of Pediatric Neuro-Oncology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAS2936
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Pontine and Thalamic Gliomas; Diffuse Midline Glioma
Keywords: Blood brain barrier; Diffuse Midline Gliomas; Convection-Enhanced Delivery (CED); Diffuse Intrinsic Pontine Glioma; Thalamic Gliomas
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- MTX110 and CED (Experimental): All patients enrolled in the study will receive infusion of MTX110 and Gadolinium delivered by the CED delivery system directly into the tumor over 9-11 days.
  Interventions: Drug: Infusate with MTX110 and gadolinium; Device: Convection-Enhanced Delivery (CED)

INTERVENTIONS:
Drug: Infusate with MTX110 and gadolinium — Pulses 1 and 2 will be prepared with 30, 60 or 90 uM concentration of MTX110. The infusate consists of gadolinium and MTX110 (30, 60, or 90 uM) at approximately 1:100 ratio.
Device: Convection-Enhanced Delivery (CED) — CED is the method by which the drug are delivered to the brain under controlled pressure to the brain by targeted micro-catheters.

SUMMARY:
The blood brain barrier (BBB) prevents some drugs from successfully reaching the target source. Convection-Enhanced Delivery (CED) is a method of direct infusion of drugs under controlled pressure to the tumor that may reduce systemic side effects of drugs in the patient.

The purpose of this Phase I study is to find the maximum tolerated dose of MTX110 (a water-soluble Panobinostat nanoparticle formulation) and Gadolinium that can be given safely in children with newly diagnosed diffuse midline gliomas. All patients enrolled in the study will receive infusion of MTX110 and Gadolinium delivered with a pump directly into the tumor over 9-11 days.

DETAILED DESCRIPTION:
Diffuse midline gliomas (DMGs), constitute 10% of all pediatric central nervous system (CNS) tumors. Subjects with Diffuse Intrinsic Pontine Gliomas (DIPG) have a poor prognosis with a median survival that is usually reported to be 9 months, and nearly 90% of children die within 18 months from diagnosis. The mainstay of treatment is radiation to the primary tumor site. Surgical resection does not influence outcome and is often not feasible in this part of the central nervous system.

Many promising drugs for central nervous system (CNS) disorders have failed to attain clinical success due to an intact blood brain barrier (BBB), limiting their access form the systemic circulation into the brain. Systemic administration of high doses may increase delivery to the brain, but this approach risks significant side effects and systemic toxicities. Direct delivery of the drugs to the brain by injection into the parenchyma bypasses the BBB, however, drug distribution form the site of injection tends to be limited. The convection-enhanced delivery (CED) of drugs describes the infusion of drugs under controlled pressure to the brain parenchyma via targeted microcatheter. This technique facilitates and deliver higher drug concentrations in brain tissue or tumor. The BBB can now operate to retain drug and to significantly reduce systemic side effects. In addition, the fact that panobinostat seems to be most efficacious clinically available drug against DIPG cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 3 years up to the 18th birthday
* Radiological diagnosis of DIPG with tumor confined to the region of the pons or
* thalami without cystic changes or hematoma obstructing the planned catheter trajectories
* Radiological diagnosis of thalamic gliomas confined to bilateral thalami without cystic changes or hematoma obstructing the planned catheter trajectories
* Radiological features of DIPG: intrinsic, pontine based infiltrative lesion; hypointense in T1 weighted images (T1WIs) and hyperintense in T2 sequences, with mass effect on the adjacent structures and occupying at least 50% of the pons
* No prior therapy is allowed other than involved field radiotherapy (54Gy) and cerebrospinal fluid (CSF) diversion for hydrocephalus, including endoscopic third ventriculostomy (ETV) or a ventriculo-peritoneal shunt. No concomitant medicine or therapies for treatment are permitted while the patient is enrolled in this study.
* Karnofsky performance status or Lansky play score of ≥70 assessed at diagnosis
* Total bilirubin: within normal institutional limits
* Aspartate Aminotransferase (AST)(SGOT)/Alanine Aminotransferase (ALT)(SGPT): ≤ 2.5 × institutional upper limit of normal (ULN)
* Creatinine: within normal institutional limits
* Creatinine clearance: ≥ 60 mL/min/1.73m2 for patients with creatinine levels above institutional normal
* Absolute neutrophil count: ≥ 1,500/μL
* Platelet count: ≥ 100,000/μL - no transfusion within 7 days
* Hemoglobin level: ≥ 10g/dL - no transfusion within 7 days
* Partial Thromboplastin Time (PT) and activated partial thromboplastin time (APTT): within normal institutional limits
* No documented current bleeding disorder
* No medical condition that would preclude general anesthesia
* No severe acute infection or unexplained febrile illness
* Not pregnant or nursing - negative serum pregnancy test if appropriate within 7 days of study entry (adequate contraceptive methods for females and males required)
* No documented allergy to compounds of similar chemical or biologic composition to MTX110 or gadolinium compounds
* Subjects with a history of seizures/epilepsy should be on anticonvulsant medication prior to the first operative procedure on study, with serum levels within a therapeutic range
* Subjects must be able to undergo MR-imaging with gadolinium-based contrast administration (e.g. no ferrous-containing implants, no pacemakers, etc.)
* All subjects or their legal guardians must sign a document of informed consent indicating their understanding of the investigational nature and the potential risks associated with this study. When appropriate, pediatric subjects will be included in all discussions in order to obtain verbal and written assent

Exclusion Criteria:

* Radiological evidence of distant disease outside the pons or thalami
* Radiological evidence of metastatic disease within the central nervous system (CNS) at diagnosis
* Subjects with an uncorrectable bleeding disorder
* Subjects with multifocal or leptomeningeal disease beyond the pons or the thalami
* Subjects with signs of impending herniation or an acute intratumoral hemorrhage
* Subjects that have received or are on concurrent chemotherapy or biologic therapy for the treatment of their tumor
* Subjects who are pregnant or breastfeeding
* Previous experimental or trial-based therapy
* Patients who are known human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C positive. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with MTX110.
* Patients with systemic diseases which may be associated with unacceptable anesthetic/operative risk

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to six weeks after second infusion
  Safety of repeated convection-enhanced delivery (CED) of MTX110 will be reported by summarizing the incidence rate of adverse events observed or reported. Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Maximum Tolerated Dose (MTD) of MTX110 | 14 days
  The MTD will be determined based on the number of dose limiting toxicities (DLT) observed in each of the titrated doses.

SECONDARY OUTCOMES:
Steady state volume of drug distribution | 14 days
  Measured by volumetric contrast enhancement intensity on MRI and magnetic resonance (MR) spectroscopy
Time to tumor progression/recurrence (PFS) | 2 years
  PFS is defined as the duration of time from start of MTX110 treatment to time of progression or death from any cause, whichever occurs first.
Overall survival (OS) or time to death | 2 years
  Overall survival is defined as the duration of time from the start of MTX110 treatment to death from any cause. OS will be measured by follow-up with a study participant every 3-6 months until death for any reason.
Score on PedsQL 4.0 Brain Tumor Module | 2 years
  The 24-item PedsQL 4.0 Brain Tumor Module encompasses six scales: (1) cognitive problems (seven items), (2) pain and hurt (three items), (3) movement and balance (three items), (4) procedural anxiety (three items), (5) nausea (five items), and (6) worry (three items). Each item is measured with a 5-point Likert scale from 0 (never a problem) to 4 (almost always a problem), which is then transformed on a scale from 0-100. Higher scores indicate lower problems and therefore a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Szalontay, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No